CLINICAL TRIAL: NCT02777554
Title: A Phase 1, Open Label, Randomized, Two Part Study to Evaluate the Pharmacokinetic Exposure of a Once-Daily (QD) Apremilast Formulation Relative to the Twice-Daily (BID) Reference Immediate Release (IR) Tablet and the Effect of Food on the QD Apremilast Formulation in Healthy Subjects.
Brief Title: A Study to Evaluate the Pharmacokinetic Exposure of 2 Formulations of Apremilast in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CC-10004-CP-035
Expanded Access: NCT03740516 (No longer available)
Record Dates: First submitted 2016-05-11; First posted 2016-05-19 (Estimated); Results first posted 2021-07-22 (Actual); Last update posted 2021-07-22 (Actual); Status verified 2021-06

CONDITIONS: Healthy Volunteers
Keywords: Healthy Subjects; Apremilast; Pharmacokinetic
MeSH Terms: interventions — apremilast

ARMS (6):
- Part 1: Apremilast 30 mg IR BID / Apremilast 75 mg XL QD (Experimental): Participants received apremilast 30 mg immediate release (IR) tablet twice a day (BID) for 7 days in treatment period 1 then apremilast 75 mg extended release (XL) formulation once a day (QD) for 7 days in treatment period 2.
  Interventions: Drug: Apremilast IR; Drug: Apremilast XL
- Part 1: Apremilast 75 mg XL QD / Apremilast 30 mg IR BID (Experimental): Participants received apremilast 75 mg XL formulation once a day for 7 days in treatment period 1 then apremilast 30 mg IR tablet twice a day for 7 days in treatment period 2.
  Interventions: Drug: Apremilast IR; Drug: Apremilast XL
- Part 2: Sequence 1 (Experimental): Participants received a single dose of apremilast in each of 4 treatment periods according to the following:
  Treatment period 1: Apremilast 30 mg IR tablet under fasted conditions; Treatment period 2: Apremilast 75 mg XL formulation after a high-fat meal; Treatment period 3: Apremilast 75 mg XL formulation under fasted conditions; Treatment period 4: Apremilast 75 mg XL formulation after a standard meal.
  Interventions: Drug: Apremilast IR; Drug: Apremilast XL
- Part 2: Sequence 2 (Experimental): Participants received a single dose of apremilast in each of 4 treatment periods according to the following:
  Treatment period 1: Apremilast 75 mg XL formulation under fasted conditions; Treatment period 2: Apremilast 30 mg IR tablet under fasted conditions; Treatment period 3: Apremilast 75 mg XL formulation after a standard meal; Treatment period 4: Apremilast 75 mg XL formulation after a high-fat meal.
  Interventions: Drug: Apremilast IR; Drug: Apremilast XL
- Part 2: Sequence 3 (Experimental): Participants received a single dose of apremilast in each of 4 treatment periods according to the following:
  Treatment period 1: Apremilast 75 mg XL formulation after a standard meal; Treatment period 2: Apremilast 75 mg XL formulation under fasted conditions; Treatment period 3: Apremilast 75 mg XL formulation after a high-fat meal; Treatment period 4: Apremilast 30 mg IR tablet under fasted conditions.
  Interventions: Drug: Apremilast IR; Drug: Apremilast XL
- Part 2: Sequence 4 (Experimental): Participants received a single dose of apremilast in each of 4 treatment periods according to the following:
  Treatment period 1: Apremilast 75 mg XL formulation after a high-fat meal; Treatment period 2: Apremilast 75 mg XL formulation after a standard meal; Treatment period 3: Apremilast 30 mg IR tablet under fasted conditions; Treatment period 4: Apremilast 75 mg XL formulation under fasted conditions.
  Interventions: Drug: Apremilast IR; Drug: Apremilast XL

INTERVENTIONS:
Drug: Apremilast IR — Apremilast immediate release tablet
  Other Names: Otezla®
Drug: Apremilast XL — Apremilast extended release formulation tablet

SUMMARY:
The purpose of this study is to evaluate the relative bioavailability of apremilast once-daily formulation relative to a twice daily formulation when administered as multiple doses (Part 1), and when administered as a single dose under fasting and fed conditions (Part 2). Information on safety and tolerability will also be obtained.

DETAILED DESCRIPTION:
Part 1: This is an open-label, randomized, two-period, two-sequence, crossover study in healthy subjects. The study will consist of a screening phase, a baseline phase, two treatment periods, and a follow-up phone call. Each period will be ten days in duration including 7 days of dosing and sample collection for up to 72 hours post Day 7 morning dose. There will be a washout between period 1 and period 2.

Part 2: This is an open-label, randomized, four-period, four-sequence crossover study to evaluate the PK and exposure of apremilast following single dose administration of different formulations of apremilast. Part 2 will consist of a screening phase, baseline, four treatment periods, and a follow-up phone call. Each period will be four days in duration for dosing (Day 1) and sample collection for up to 72 hours post Day 1.

ELIGIBILITY:
Inclusion Criteria:

Subjects must satisfy the following criteria to be enrolled in the study (Part 1 and Part 2):

1. Must understand and voluntarily sign a written Informed consent form (ICF) prior to any study-related procedures being performed.
2. Must be able to communicate with the investigator, understand and comply with the requirements of the study, and agree to adhere to restrictions and examination schedules.
3. Male and female subjects of any race between 18 to 55 years of age (inclusive), and in good health as determined by the Investigator at the time of signing the informed consent document.
4. Have a body mass index (BMI) between 18 and 33 kg/m^2 (inclusive).
5. No clinically significant laboratory test results as determined by the investigator.
6. At the screening visit, must be afebrile, with supine systolic blood pressure (BP): 90 to 140 mmHg, supine diastolic BP: 50 to 90 mmHg, and pulse rate: 40 to 110 bpm. Eligibility criteria for vital signs performed during check-in and/or predose on Day 1 will be at the discretion of the Investigator.
7. Must have a normal or clinically acceptable 12-lead electrocardiogram (ECG). Subjects must have a QT interval corrected using the Fridericia formula (QTcF) value ≤ 450 msec.
8. Female subjects

   1. Must have a negative pregnancy test
   2. If postmenopausal: must have follicular stimulating hormone (FSH) test result > 40 IU/L and a negative pregnancy test
9. Contraception Requirements:

   Must comply with the following acceptable forms of contraception. All Female of child bearing potential (FCBP)1 must use one of the approved contraceptive options as described below while taking apremilast and for at least 28 days after administration of the last dose of the apremilast. At the time of study entry, and at any time during the study when a FCBP's contraceptive measures or ability to become pregnant changes, the Investigator will educate the subject regarding contraception options and the correct and consistent use of effective contraceptive methods in order to successfully prevent pregnancy.

   All FCBP must have a negative pregnancy test at Screening and Day -1 of each Treatment Period. All FCBP subjects who engage in activity in which conception is possible must use one of the approved contraceptive options described below:

   Option 1: Any one of the following highly effective methods: hormonal contraception (oral, injection, implant, transdermal patch, vaginal ring); intrauterine device (IUD); tubal ligation; or partner's vasectomy; OR Option 2: Male or female condom (latex condom or non-latex condom NOT made out of natural [animal] membrane [for example, polyurethane]); Plus one additional barrier(c) contraceptive sponge with spermicide.

   Male subjects (including those who have had a vasectomy) who engage in activity in which conception is possible must use barrier contraception (latex or non-latex condoms NOT made out of natural [animal] membrane [for example, polyurethane]) while on Investigational Product (IP) and for at least 28 days after the last dose of IP.
10. Must agree to refrain from donating sperm, blood or plasma (other than for this study) while participating in this study and for at least 28 days after the last dose of investigational product.
11. Subject is willing and able to adhere to the study visit schedule and other protocol requirements.

Exclusion Criteria:

The presence of any of the following will exclude a subject from enrollment:

1. History of any clinically significant and relevant neurological, psychiatric, gastrointestinal, renal, hepatic, cardiovascular, psychological, pulmonary, metabolic, endocrine, hematological, allergic disease, drug allergies, or other major disorders.
2. Any condition which places the subject at unacceptable risk if he were to participate in the study, or confounds the ability to interpret data from the study.

1 A female of childbearing potential is a sexually mature female who 1) has not undergone a hysterectomy (the surgical removal of the uterus) or bilateral oophorectomy (the surgical removal of both ovaries) or 2) has not been postmenopausal for at least 24 consecutive months (that is, has had menses at any time during the preceding 24 consecutive months).

3. Use of any prescribed systemic or topical medication within 30 days of the first dose administration (exception, FCBP may use hormonal contraception).

4. Use of any non-prescribed systemic or topical medication (including vitamin/mineral supplements, and herbal medicines) within 14 days of the first dose administration.

5. Any surgical or medical condition possibly affecting drug absorption, distribution, metabolism and excretion, eg, bariatric procedure, colon resection, irritable bowel syndrome, Crohn's disease, etc. Subjects with cholecystectomy and appendectomy may be included.

6. Exposure to an investigational drug (new chemical entity) within 30 days prior to the first dose administration or 5 half-lives of that investigational drug, if known (whichever is longer).

7. Donated blood or plasma within 8 weeks before the first dose administration to a blood bank or blood donation center.

8. History of drug abuse (as defined by the current version of the Diagnostic and Statistical Manual [DSM]) within 2 years before dosing, or a positive drug screen reflecting consumption of illicit drugs.

9. History of alcohol abuse (as defined by the current version of the DSM) within 2 years before dosing, or a positive alcohol screen.

10. Known to have hepatitis, or known to be a carrier of the hepatitis B surface antigen (HBsAg) or hepatitis C antibody (HCV Ab), or have a positive result to the test for human immunodeficiency virus (HIV) antibodies at screening.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 144 (Actual)
Dates: Start 2016-08-17 (Actual); Primary Completion 2016-11-22 (Actual); Study Completion 2016-11-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (2):
- United States (2):
  - Covance-Daytona Beach, Daytona Beach, Florida
  - Covance Clinical Research Unit Inc, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: http://www.amgen.com/datasharing

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 2 clinical sites in the United States. The study consisted of 2 parts. Part 1 was a multiple-dose two-period, two-sequence, crossover study. Part 2 was a four-period, four-sequence crossover study. Both parts enrolled healthy volunteers.
Pre-assignment Details: In Part 1 participants were randomly assigned to 1 of 2 treatment sequences. In Part 2 participants were randomly assigned to 1 of 4 treatment sequences.
Groups:
- Part 1: Apremilast 30 mg IR BID / Apremilast 75 mg XL QD: Participants received apremilast 30 mg immediate release (IR) tablet twice a day (BID) for 7 days in treatment period 1 then apremilast 75 mg extended release (XL) formulation once a day (QD) for 7 days in treatment period 2. There was a 5.5 to 9.5-day washout period between each treatment period.
- Part 1: Apremilast 75 mg XL QD / Apremilast 30 mg IR BID: Participants received apremilast 75 mg XL formulation once a day for 7 days in treatment period 1 then apremilast 30 mg IR tablet twice a day for 7 days in treatment period 2. There was a 6 to 10-day washout period between each treatment period.
- Part 2: Sequence 1: Participants received a single dose of apremilast in each of 4 treatment periods according to the following:
  Treatment period 1: Apremilast 30 mg IR tablet in the morning and evening under fasted conditions; Treatment period 2: Apremilast 75 mg XL formulation after a high-fat meal; Treatment period 3: Apremilast 75 mg XL formulation under fasted conditions; Treatment period 4: Apremilast 75 mg XL formulation after a standard meal. There was a washout period of approximately 6 to 10 days between each treatment period.
- Part 2: Sequence 2: Participants received a single dose of apremilast in each of 4 treatment periods according to the following:
  Treatment period 1: Apremilast 75 mg XL formulation under fasted conditions; Treatment period 2: Apremilast 30 mg IR tablet in the morning and evening under fasted conditions; Treatment period 3: Apremilast 75 mg XL formulation after a standard meal; Treatment period 4: Apremilast 75 mg XL formulation after a high-fat meal. There was a washout period of approximately 6 to 10 days between each treatment period.
- Part 2: Sequence 3: Participants received a single dose of apremilast in each of 4 treatment periods according to the following:
  Treatment period 1: Apremilast 75 mg XL formulation after a standard meal; Treatment period 2: Apremilast 75 mg XL formulation under fasted conditions; Treatment period 3: Apremilast 75 mg XL formulation after a high-fat meal; Treatment period 4: Apremilast 30 mg IR tablet in the morning and evening under fasted conditions.
  There was a washout period of approximately 6 to 10 days between each treatment period.
- Part 2: Sequence 4: Participants received a single dose of apremilast in each of 4 treatment periods according to the following:
  Treatment period 1: Apremilast 75 mg XL formulation after a high-fat meal; Treatment period 2: Apremilast 75 mg XL formulation after a standard meal; Treatment period 3: Apremilast 30 mg IR tablet in the morning and evening under fasted conditions; Treatment period 4: Apremilast 75 mg XL formulation under fasted conditions. There was a washout period of approximately 6 to 10 days between each treatment period.
Period: Overall Study
Arm/Group | Part 1: Apremilast 30 mg IR BID / Apremilast 75 mg XL QD | Part 1: Apremilast 75 mg XL QD / Apremilast 30 mg IR BID | Part 2: Sequence 1 | Part 2: Sequence 2 | Part 2: Sequence 3 | Part 2: Sequence 4
Started | 62 | 62 | 5 | 5 | 5 | 5
Completed | 32 | 37 | 4 | 4 | 5 | 5
Not Completed | 30 | 25 | 1 | 1 | 0 | 0
Not completed — Adverse Event | 4 | 4 | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 3 | 1 | 1 | 0 | 0 | 0
Not completed — Discharged early due to hurricane | 22 | 20 | 0 | 0 | 0 | 0
Not completed — Other - Miscellaneous | 1 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All enrolled participants
Groups:
- Part 1: Participants in Part 1 received apremilast 30 mg IR tablet BID for 7 days and apremilast 75 mg XL formulation QD for 7 days in each treatment period depending on sequence assignment.
- Part 2: Participants in Part 2 received a single dose of the following treatments in 4 treatment periods according to sequence assignment:
  * Apremilast 30 mg IR tablet in the morning and evening under fasted conditions;
  * Apremilast 75 mg XL formulation after a high-fat meal;
  * Apremilast 75 mg XL formulation under fasted conditions;
  * Apremilast 75 mg XL formulation after a standard meal.
- Total: Total of all reporting groups
Arm/Group | Part 1 | Part 2 | Total
Number analyzed (Participants) | 124 | 20 | 144
Age, Continuous [Mean (Full Range); unit: years] | 37.8 [19 to 55] | 34.7 [20 to 53] | 37.4 [19 to 55]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46 | 7 | 53
  Male | 78 | 13 | 91
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 52 | 8 | 60
  Not Hispanic or Latino | 72 | 12 | 84
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Black or African American | 47 | 10 | 57
  White | 70 | 10 | 80
  Asian | 4 | 0 | 4
  Other | 2 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Part 1: Peak Maximum Plasma Concentration (Cmax) of Apremilast
Time Frame: Apremilast IR: Day 7 predose and at 0.5, 1, 2, 3, 5, 8, 12, 12.5, 13, 14, 15, 17, 20, and 24 hours after the morning dose. Apremilast XL: Day 7 predose and at 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 14, 16, 20, and 24 hours after the morning dose.
Population: The pharmacokinetic (PK) population (all participants who received at least one dose of apremilast and had at least one measurable concentration datum) with available data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- Part 1: Apremilast 30 mg IR BID: Participants received apremilast 30 mg IR tablet BID for 7 days.
- Part 1: Apremilast 75 mg XL QD: Participants received apremilast 75 mg XL formulation QD for 7 days.
Arm/Group | Part 1: Apremilast 30 mg IR BID | Part 1: Apremilast 75 mg XL QD
Number analyzed (Participants) | 91 | 89
ng/mL | 451 (49.0) | 459 (35.0)
Statistical Analysis 1: Comparison: Part 1: Apremilast 30 mg IR BID vs Part 1: Apremilast 75 mg XL QD; To assess the exposure between the extended release apremilast formulation, and Reference IR (30 mg reference IR BID) tablet following multiple oral doses, an analysis of variance (ANOVA) model, with sequence, period, and treatment as fixed effects, and subject nested within sequence as a random effect, was performed on the natural log-transformed Day 7 Cmax; Test type: Equivalence — Equivalent exposure of the QD formulation to the BID tablet was established if the 90% confidence intervals (CIs) of the geometric mean ratio for Day 7 AUC0-24 and Cmax were completely contained within the range of 80% to 125%; Ratio (%) of Geometric Means = 101.6, 90% CI 2-sided [95.1 to 108.5] — Geometric mean ratio (Apremilast 75 mg XL QD / Apremilast 30 mg IR BID) from an ANOVA model, expressed as a percentage

2. Primary Outcome: Part 1: Area Under the Concentration-time Curve From Time Zero to 24 Hours Postdose (AUC0-24) of Apremilast
Time Frame: as for outcome 1
Population: The PK population with available data
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Part 1: Apremilast 30 mg IR BID | Part 1: Apremilast 75 mg XL QD
Number analyzed (Participants) | 91 | 89
ng*hr/mL | 6370 (51.2) | 6090 (46.1)
Statistical Analysis 1: Comparison: Part 1: Apremilast 30 mg IR BID vs Part 1: Apremilast 75 mg XL QD; To assess the exposure between the extended release apremilast formulation, and Reference IR (30 mg reference IR BID) tablet following multiple oral doses, an ANOVA model, with sequence, period, and treatment as fixed effects, and subject nested within sequence as a random effect, was performed on the natural log-transformed Day 7 AUC0-24; Test type: Equivalence — Equivalent exposure of the QD formulation to the BID tablet was established if the 90% CIs of the geometric mean ratio for Day 7 AUC0-24 and Cmax were completely contained within the range of 80% to 125%; Ratio (%) of Geometric Means = 95.3, 90% CI 2-sided [88.9 to 102.2] — Geometric mean ratio (Apremilast 75 mg XL QD / Apremilast 30 mg IR BID) from an ANOVA model, expressed as a percentage

3. Primary Outcome: Part 2: Peak Maximum Plasma Concentration (Cmax) of Apremilast
Time Frame: Apremilast IR: Predose and at 0.5, 1, 2, 3, 5, 8, 12, 12.5, 13, 14, 15, 17, 20, 24, 36, 48, 60, and 72 hours after the morning dose. Apremilast XL: Predose and at 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 14, 16, 20, 24, 30, 36, 48, 60, and 72 hours postdose.
Population: PK population; two participants were excluded from PK analyses due to predose concentrations > 5% than their Cmax values.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- Part 2: Apremilast 30 mg IR BID (Fasted): Participants received one apremilast 30 mg IR tablet in the morning and one in the evening under fasted conditions.
- Part 2: Apremilast 75 mg XL (Fasted): Participants received a single dose of apremilast 75 mg XL formulation under fasted conditions.
- Part 2: Apremilast 75 mg XL (Standard Meal): Participants received a single dose of apremilast 75 mg XL formulation after a standard meal.
- Part 2: Apremilast 75 mg XL (High Fat Meal): Participants received a single dose of apremilast 75 mg XL formulation after a high-fat meal.
Arm/Group | Part 2: Apremilast 30 mg IR BID (Fasted) | Part 2: Apremilast 75 mg XL (Fasted) | Part 2: Apremilast 75 mg XL (Standard Meal) | Part 2: Apremilast 75 mg XL (High Fat Meal)
Number analyzed (Participants) | 18 | 17 | 16 | 17
ng/mL | 379 (29.9) | 402 (32.5) | 436 (33.2) | 496 (25.2)
Statistical Analysis 1: Comparison: Part 2: Apremilast 30 mg IR BID (Fasted) vs Part 2: Apremilast 75 mg XL (Fasted); To estimate the exposure of apremilast following single dose administration of extended release (QD) relative to the Reference IR (BID) tablet under fasted conditions, an ANOVA model with treatment, sequence, and period as fixed effects, and subject nested within sequence as a random effect, was performed on the natural log-transformed Cmax of apremilast; Test type: Other; Ratio (%) of Geometric Means = 103.9, 90% CI 2-sided [93.6 to 115.4] — Geometric mean ratio (Apremilast 75 mg XL / Apremilast 30 mg IR BID) from an ANOVA model, expressed as a percentage
Statistical Analysis 2: Comparison: Part 2: Apremilast 75 mg XL (Fasted) vs Part 2: Apremilast 75 mg XL (Standard Meal); To estimate the effect of food on the PK of a single oral dose of extended release apremilast (QD), an ANOVA model with treatment, sequence, and period as fixed effects, and subject nested within sequence as a random effect, was performed on the natural log-transformed Cmax of apremilast; Test type: Other; Ratio (%) of Geometric Means = 90.9, 90% CI 2-sided [81.6 to 101.3] — Geometric mean ratio (Apremilast 75 mg XL (Fasted) / Apremilast 75 mg XL (Standard Meal)) from an ANOVA model, expressed as a percentage
Statistical Analysis 3: Comparison: Part 2: Apremilast 75 mg XL (Standard Meal) vs Part 2: Apremilast 75 mg XL (High Fat Meal); [analysis description as in outcome 3, analysis 2]; Test type: Other; Ratio (%) of Geometric Means = 115.0, 90% CI 2-sided [103.3 to 128.1] — Geometric mean ratio (Apremilast 75 mg XL (High Fat) / Apremilast 75 mg XL (Standard Meal)) from an ANOVA model, expressed as a percentage
Statistical Analysis 4: Comparison: Part 2: Apremilast 75 mg XL (Fasted) vs Part 2: Apremilast 75 mg XL (High Fat Meal); [analysis description as in outcome 3, analysis 2]; Test type: Other; Ratio (%) of Geometric Means = 126.5, 90% CI 2-sided [113.7 to 140.8] — Geometric mean ratio (Apremilast 75 mg XL (High Fat) / Apremilast 75 mg XL (Fasted)) from an ANOVA model, expressed as a percentage

4. Primary Outcome: Part 2: Area Under the Plasma Concentration-time Curve From Time Zero to the Last Observable Concentration (AUC0-t) of Apremilast
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Part 2: Apremilast 30 mg IR BID (Fasted) | Part 2: Apremilast 75 mg XL (Fasted) | Part 2: Apremilast 75 mg XL (Standard Meal) | Part 2: Apremilast 75 mg XL (High Fat Meal)
Number analyzed (Participants) | 18 | 17 | 16 | 17
ng*h/mL | 7030 (31.5) | 6650 (42.5) | 7580 (31.1) | 7400 (31.1)
Statistical Analysis 1: Comparison: Part 2: Apremilast 30 mg IR BID (Fasted) vs Part 2: Apremilast 75 mg XL (Fasted); To estimate the exposure of apremilast following single dose administration of extended release (QD) relative to the Reference IR (BID) tablet under fasted conditions, an ANOVA model with treatment, sequence, and period as fixed effects, and subject nested within sequence as a random effect, was performed on the natural log-transformed AUC0-t of apremilast; Test type: Other; Ratio (%) of Geometric Means = 92.9, 90% CI 2-sided [81.3 to 106.2] — Geometric mean ratio (Apremilast 75 mg XL / Apremilast 30 mg IR BID) from an ANOVA model, expressed as a percentage
Statistical Analysis 2: Comparison: Part 2: Apremilast 75 mg XL (Fasted) vs Part 2: Apremilast 75 mg XL (Standard Meal); To estimate the effect of food on the PK of a single oral dose of extended release apremilast (QD), an ANOVA model with treatment, sequence, and period as fixed effects, and subject nested within sequence as a random effect, was performed on the natural log-transformed AUC0-t of apremilast; Test type: Other; Ratio (%) of Geometric Means = 86.0, 90% CI 2-sided [74.9 to 98.7] — [estimate comment as in outcome 3, analysis 2]
Statistical Analysis 3: Comparison: Part 2: Apremilast 75 mg XL (Standard Meal) vs Part 2: Apremilast 75 mg XL (High Fat Meal); [analysis description as in outcome 4, analysis 2]; Test type: Other; Ratio (%) of Geometric Means = 97.3, 90% CI 2-sided [84.9 to 111.6] — [estimate comment as in outcome 3, analysis 3]
Statistical Analysis 4: Comparison: Part 2: Apremilast 75 mg XL (Fasted) vs Part 2: Apremilast 75 mg XL (High Fat Meal); [analysis description as in outcome 4, analysis 2]; Test type: Other; Ratio (%) of Geometric Means = 113.2, 90% CI 2-sided [98.8 to 129.7] — [estimate comment as in outcome 3, analysis 4]

5. Primary Outcome: Part 2: Area Under the Plasma Concentration-time Curve From Time Zero Extrapolated to Infinity (AUC0-∞) of Apremilast
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Part 2: Apremilast 30 mg IR BID (Fasted) | Part 2: Apremilast 75 mg XL (Fasted) | Part 2: Apremilast 75 mg XL (Standard Meal) | Part 2: Apremilast 75 mg XL (High Fat Meal)
Number analyzed (Participants) | 18 | 17 | 16 | 17
ng*h/mL | 7100 (31.4) | 6680 (42.4) | 7600 (31.1) | 7450 (31.1)
Statistical Analysis 1: Comparison: Part 2: Apremilast 30 mg IR BID (Fasted) vs Part 2: Apremilast 75 mg XL (Fasted); To estimate the exposure of apremilast following single dose administration of extended release (QD) relative to the Reference IR (BID) tablet under fasted conditions, an ANOVA model with treatment, sequence, and period as fixed effects, and subject nested within sequence as a random effect, was performed on the natural log-transformed AUC0-∞ of apremilast; Test type: Other; Ratio (%) of Geometric Means = 92.6, 90% CI 2-sided [81.1 to 105.9] — Geometric mean ratio (Apremilast 75 mg XL / Apremilast 30 mg IR BID) from an ANOVA model, expressed as a percentage
Statistical Analysis 2: Comparison: Part 2: Apremilast 75 mg XL (Fasted) vs Part 2: Apremilast 75 mg XL (Standard Meal); To estimate the effect of food on the PK of a single oral dose of extended release apremilast (QD), an ANOVA model with treatment, sequence, and period as fixed effects, and subject nested within sequence as a random effect, was performed on the natural log-transformed AUC0-∞ of apremilast; Test type: Other; Ratio (%) of Geometric Means = 86.1, 90% CI 2-sided [75.0 to 98.8] — [estimate comment as in outcome 3, analysis 2]
Statistical Analysis 3: Comparison: Part 2: Apremilast 75 mg XL (Standard Meal) vs Part 2: Apremilast 75 mg XL (High Fat Meal); [analysis description as in outcome 5, analysis 2]; Test type: Other; Ratio (%) of Geometric Means = 97.5, 90% CI 2-sided [85.0 to 111.8] — [estimate comment as in outcome 3, analysis 3]
Statistical Analysis 4: Comparison: Part 2: Apremilast 75 mg XL (Fasted) vs Part 2: Apremilast 75 mg XL (High Fat Meal); [analysis description as in outcome 5, analysis 2]; Test type: Other; Ratio (%) of Geometric Means = 113.2, 90% CI 2-sided [98.8 to 129.7] — [estimate comment as in outcome 3, analysis 4]

6. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events
Description: An adverse event (AE) is any noxious, unintended, or untoward medical occurrence that may appear or worsen in a participant during the course of a study. It may be a new intercurrent illness, a worsening concomitant illness, an injury, or any concomitant impairment of the subject's health, including laboratory test values, regardless of etiology.
  A serious AE is any AE occurring at any dose that:
  * Resulted in death;
  * Was life-threatening;
  * Required inpatient hospitalization or prolongation of existing hospitalization;
  * Resulted in persistent or significant disability/incapacity;
  * Was a congenital anomaly/birth defect;
  * Constituted an important medical event. The Investigator determined the relationship between the administration of study drug and the occurrence of each AE as Not Suspected or Suspected as defined in the Protocol.
Time Frame: Part 1: Up to 7 days after last dose in each treatment period (14 days); Part 2: Up to 7 days after each dose.
Population: All participants who received at least one dose of apremilast
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Apremilast 30 mg IR BID | Part 1: Apremilast 75 mg XL QD | Part 2: Apremilast 30 mg IR BID (Fasted) | Part 2: Apremilast 75 mg XL (Fasted) | Part 2: Apremilast 75 mg XL (Standard Meal) | Part 2: Apremilast 75 mg XL (High Fat Meal)
Number analyzed (Participants) | 108 | 107 | 20 | 19 | 18 | 19
Participants
  Any treatment-emergent adverse event (TEAE) | 50 | 47 | 2 | 4 | 3 | 2
  TEAE related to study drug | 45 | 41 | 2 | 3 | 2 | 2
  Serious adverse events | 0 | 0 | 0 | 0 | 0 | 0
  Serious adverse events related to study drug | 0 | 0 | 0 | 0 | 0 | 0
  TEAE leading to discontinuation | 3 | 5 | 1 | 0 | 0 | 0
  TEAE related to study drug leading to discontinuation | 3 | 5 | 1 | 0 | 0 | 0
  Deaths | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Part 1: Up to 7 days after last dose in each treatment period (14 days); Part 2: Up to 7 days after each dose.
Groups:
- Part 1 Total: Participants in Part 1 received apremilast 30 mg IR tablet BID for 7 days and apremilast 75 mg XL formulation QD for 7 days in each treatment period depending on sequence assignment.
- Part 2: Apremilast 30 mg IR (Fasted): Participants received one apremilast 30 mg IR tablet in the morning and one in the evening under fasted conditions
- Part 2 Total: Participants in Part 2 received a single dose of the following treatments in 4 treatment periods according to sequence assignment:
  * Apremilast 30 mg IR tablet in the morning and evening under fasted conditions;
  * Apremilast 75 mg XL formulation under fasted conditions;
  * Apremilast 75 mg XL formulation after a standard meal;
  * Apremilast 75 mg XL formulation after a high-fat meal.
Arm/Group | Part 1: Apremilast 30 mg IR BID | Part 1: Apremilast 75 mg XL QD | Part 1 Total | Part 2: Apremilast 30 mg IR (Fasted) | Part 2: Apremilast 75 mg XL (Fasted) | Part 2: Apremilast 75 mg XL (Standard Meal) | Part 2: Apremilast 75 mg XL (High Fat Meal) | Part 2 Total
Serious Adverse Events (participants affected / at risk) | 0/108 | 0/107 | 0/124 | 0/20 | 0/19 | 0/18 | 0/19 | 0/20
Other Adverse Events (participants affected / at risk) | 41/108 | 35/107 | 59/124 | 2/20 | 4/19 | 3/18 | 2/19 | 8/20
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: Apremilast 30 mg IR BID (N=108) | Part 1: Apremilast 75 mg XL QD (N=107) | Part 1 Total (N=124) | Part 2: Apremilast 30 mg IR (Fasted) (N=20) | Part 2: Apremilast 75 mg XL (Fasted) (N=19) | Part 2: Apremilast 75 mg XL (Standard Meal) (N=18) | Part 2: Apremilast 75 mg XL (High Fat Meal) (N=19) | Part 2 Total (N=20)
Abdominal pain (Gastrointestinal disorders) | 4 | 3 | 6 | 1 | 1 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 15 | 13 | 21 | 1 | 2 | 0 | 0 | 2
Dyspepsia (Gastrointestinal disorders) | 3 | 0 | 3 | 1 | 0 | 1 | 0 | 1
Nausea (Gastrointestinal disorders) | 11 | 7 | 16 | 1 | 1 | 0 | 2 | 3
Vomiting (Gastrointestinal disorders) | 2 | 3 | 5 | 1 | 0 | 0 | 1 | 2
Fatigue (General disorders) | 5 | 5 | 7 | 0 | 0 | 0 | 0 | 0
Malaise (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Pain (General disorders) | 6 | 0 | 6 | 0 | 0 | 0 | 0 | 0
Hypovolaemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 7 | 8 | 0 | 0 | 0 | 0 | 0
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 6 | 3 | 8 | 0 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 8 | 8 | 15 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 2 | 2 | 4 | 1 | 1 | 0 | 0 | 2
Headache (Nervous system disorders) | 27 | 25 | 43 | 0 | 1 | 2 | 2 | 5
Lethargy (Nervous system disorders) | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.